CLINICAL TRIAL: NCT06319690
Title: Combined Effects of Lion's Breath Technique With Chest Percussion Therapy in Pneumonia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0362
Record Dates: First submitted 2024-03-04; First posted 2024-03-20 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Pneumonia
Keywords: Breathing exercises; Lion's Breath Technique; Pulmonary rehabilitation
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial (RCT)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Lion breath) (Experimental): Lion's Breath Technique + Chest Percussion Therapy
  Interventions: Other: Lion's Breath Technique; Other: Chest Percussion Therapy
- Control Group (Routine treatment) (Active Comparator): Chest Percussion Therapy only
  Interventions: Other: Chest Percussion Therapy

INTERVENTIONS:
Other: Lion's Breath Technique — Patients receive training in Lion's Breath Technique, emphasizing deep diaphragmatic breathing and controlled exhalation.
  Daily supervised Lion's Breath Technique sessions for 20 minutes for 1 week
  Arms: Experimental Group (Lion breath)
Other: Chest Percussion Therapy — Trained physiotherapists administer chest percussion therapy to mobilize secretions and improve lung function.
  Daily session for 30 minutes for 1 week.

SUMMARY:
This study will be randomized controlled trial with non-probability convenient sampling. Sample size will be 90,45 in each group. Outcome will be measured by using 6 minute walk test, Spirometry (FVC, FEV1/FVC and PEF), Functional Independence Measure.

DETAILED DESCRIPTION:
The main objective of the study is to determine the effect of lion's breath technique along with chest percussion therapy in pneumonia patients. This study will be randomized controlled trial with non-probability convenient sampling. Sample size will be 90,45 in each group. Participants included will be adults aged 18 years and above diagnosed with pneumonia. Willing to comply with the study protocol. Both male and female will be included. Participants should be in stable health conditions to participate in the Study. Patients with severe or life-threatening pneumonia requiring immediate intensive care and patients with physical or cognitive limitations. Patients with a history of chronic respiratory conditions such as COPD, bronchitis, or asthma. Pregnant or breastfeeding women. Individuals with musculoskeletal or neurological conditions and Patients with contraindications to chest percussion therapy, such as recent surgery or trauma to the chest area will be excluded. Group A (Lion's Breath Technique + Chest Percussion Therapy) Daily supervised Lion's Breath Technique sessions will be for 20 minutes for 1 week. Trained physiotherapists administer chest percussion therapy will be to mobilize secretions and improve lung function. Daily session for 30 minutes for 1 week. Pre and post data will be gathered. Outcome will be measured by using 6 minute walk test, Spirometry (FVC, FEV1/FVC and PEF), Functional Independence Measure.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the post-acute phase of pneumonia recovery.
* Adults aged 18 years and above diagnosed with pneumonia.
* Both male and female will be included.
* Participants should be in stable health conditions to participate in the Study.
* Willing to comply with the study protocol

Exclusion Criteria:

* Patients with severe or life-threatening pneumonia requiring immediate intensive care
* Patients with physical or cognitive limitations
* Patients with a history of chronic respiratory conditions such as COPD, bronchitis, or asthma
* Pregnant or breastfeeding women
* Individuals with musculoskeletal or neurological conditions
* Patients with contraindications to chest percussion therapy, such as recent surgery or trauma to the chest area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
George respiratory questionnaire | 1 Week
  The George respiratory questionnaire is Disease-specific instrument designed to measure the impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. Total 50 items, 2 parts (3 components). Part 1 : Symptoms component (frequency & severity) with a 1, 3 or 12-month recall (best performance with 3- and 12-month recall); Part 2: Activities that cause or are limited by breathlessness; Impact components (social functioning, psychological disturbances resulting from airways disease) refer to current state as the recall.
  Part I (Symptoms): several scales; Part II (Activity and Impacts): dichotomous (true/false) except last question (4-point Likert scale) Scores range from 0 to 100, with higher scores indicating more limitations.
Forced vital capacity (FVC) | 1 Week
  Forced vital capacity (FVC) is the amount of air that can be forcibly exhaled from your lungs after taking the deepest breath possible. It's measured by spirometry
Borg Dyspnea Scale | 1 Week
  The borg dyspnea scale is a numerical scale that measures the intensity of breathlessness of fatigue. It will be used to assess the baseline and posttest symptoms of patients with respiratory and cardiac condition.
  This is a scale that asks you to rate the difficulty of your breathing. It starts at number 0 where your breathing is causing you no difficulty at all and progresses through to number 10 where your breathing difficulty is maximal
Forced expiratory volume (FEV1) | 1 Week
  Forced expiratory volume (FEV1) calculates the amount of air that a person can force out of their lungs in 1 second. it is measured using Spirometer.
FEV1/FVC Ratio | 1 Week
  The FEV1/FVC ratio is the ratio of the forced expiratory volume in the first one second to the forced vital capacity of the lungs. The normal value for this ratio is above 0.75-85, measured using Spirometer.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Faizan Hamid, MS-CPPT, Principal Investigator — Riphah International University
Locations (1):
- Jinnah Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No